CLINICAL TRIAL: NCT05766774
Title: Feeding Study to Optimize Endocrine Dysfunction in Cystic Fibrosis
Brief Title: FEED-Cystic Fibrosis (FEED-CF)
Acronym: FEED-CF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jessica Alvarez, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00004517; 1R01DK133523-01 (NIH)
Record Dates: First submitted 2023-02-21; First posted 2023-03-13 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis-related Diabetes
MeSH Terms: conditions — Cystic Fibrosis | interventions — Diet, High-Fat

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, parallel-group design clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study team, including the investigators, statistician, and coordinator, will be blinded to diet allocation throughout. All major assessments and assays will be performed by individuals who will be blinded to the diet. Participants will not be informed of their allocated diet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-added sugar, high-fat diet Arm (Experimental): Patients will receive a low-added sugar, high-fat diet for 8 weeks. Study menus will be designed by registered dietitians using the Nutrient Database System for Research (NDSR) software program with a 2-wk rotation.Total kcal provided will be individually tailored to maintain body weight and adjusted throughout as needed. All foods (including snacks and drinks) for 8 wks will be delivered to participants' homes. Menus will be designed so that food will be delivered to subjects' homes every 3-4 days. It will be expected that participants consume only the foods provided by the study.
  Interventions: Other: Low-added sugar, high-fat diet
- Typical CF diet Arm (Active Comparator): Patients will receive a high-added sugar, high-fat CF diet for 8 weeks. Study menus will be designed by registered dietitians using the Nutrient Database System for Research (NDSR) software program with a 2-wk rotation. Total kcal provided will be individually tailored to maintain body weight and adjusted throughout as needed. All foods (including snacks and drinks) for 8 wks will be delivered to participants' homes. Menus will be designed so that food will be delivered to subjects' homes every 3-4 days. It will be expected that participants consume only the foods provided by the study.
  Interventions: Other: High-added sugar, high-fat CF diet

INTERVENTIONS:
Other: Low-added sugar, high-fat diet — Consist of <5% kcal from added sugars as recommended by the American Heart Association, and the glycemic index will be 45 or lower (25% lower than typical CF diet). The macronutrient composition of both study diets will reflect the general CF recommendations for macronutrients: 35-40% of total kcal from fat and 15-20% total kcal from protein.
  Arms: Low-added sugar, high-fat diet Arm
Other: High-added sugar, high-fat CF diet — Consist of ≥13% kcal from added sugars and the glycemic index will be >60. The macronutrient composition of both study diets will reflect the general CF recommendations for macronutrients: 35-40% of total kcal from fat and 15-20% total kcal from protein.
  Other Names: Typical CF diet
  Arms: Typical CF diet Arm

SUMMARY:
The goal of this study is to determine the extent to which excess dietary sugars serve as a precipitating factor in glucose intolerance in adults with cystic fibrosis (CF), a population at especially high risk for a unique form of diabetes (CF-related diabetes, CFRD) and with standard-of-care dietary recommendations (high-calorie, high-fat) that conflict with recommendations for other forms of diabetes.

This trial will investigate if the typical high-sugar, high-fat CF diet plays a role in diabetes risk and visceral fat accumulation in people with CF. A total of 30 participants will get a low-added sugar, high-fat diet and the other 30 will get a standard CF diet with no sugar restrictions. Participants will be randomized to the diet group they are assigned. All foods will be provided for 8 weeks.

DETAILED DESCRIPTION:
Approximately half of adults with cystic fibrosis (CF), a genetic disease, will develop diabetes. Dietary strategies shown to be successful in preventing or treating other forms of diabetes in people without CF contradict current nutritional recommendations for people with CF. The nutrition standard-of-care in CF is prescription of an unrestricted high-calorie, high-fat diet because of malnutrition. However, the standard CF diet translates to low-quality diets, with excess added sugars well-above general population recommendations. Also the investigators have shown that people with CF have more fat around their abdominal organs (called visceral fat) compared to healthy controls. The hypothesis is that the typical high-sugar, high-fat CF diet plays a role in diabetes risk and visceral fat accumulation in people with CF. In this study, the investigators will test if a low-added sugar diet improves risk markers for diabetes and decreases visceral fat over 8 weeks. The study will recruit 60 participants with CF. A total of 30 participants will get a low-added sugar, high-fat diet and the other 30 will get a standard CF diet with no sugar restrictions. Participants will be randomized to the diet group they are assigned. All foods will be provided for 8 weeks. There will be a total of 4 study visits at the Emory Hospital clinical research unit. These will include: 1) a screening visit with an oral glucose tolerance test with blood draws to determine if they already have diabetes, 2) a baseline visit for an insulin secretion test (called glucose-potentiated arginine (GPA) stimulation test) to assess risk for diabetes, as well as magnetic resonance imaging (MRI) testing to measure visceral fat, 3) a 4-week visit for another oral glucose tolerance test and in-person check-in, and 4) an 8-week visit for another GPA and MRI. Blood samples will be collected and banked. In addition to all meals provided for 8 weeks, participants will be compensated for their time and effort. Participants will be recruited from patients seen at the Emory CF Clinic. Informed consent will be performed prior to any study testing. The investigators hope this study will contribute to the development of new standardized nutrition guidelines for people living with CF.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed CF diagnosis
2. Ages 18 years and older
3. Baseline estimated daily total added sugar intake >16 tsp, as estimated from the Dietary Screener Questionnaire (DSQ).

Exclusion Criteria:

1. Nocturnal tube feeds
2. BMI <18.5 kg/m2
3. Life expectancy < 12 months
4. Confirmed diagnosis of CFRD
5. Screening OGTT showing fasting hyperglycemia (≥126 mg/dL)
6. Chronic steroid use
7. Current pregnancy or lactation
8. Inability/unwillingness to consume the majority of foods on the menu during the study period
9. MRI-incompatible metal that cannot be removed for testing
10. Uncontrolled exocrine pancreatic insufficiency/malabsorption
11. Clinically instability, defined as no changes in medical regimen (including medications and pulmonary exacerbations) for at least 21 days prior to study visit
12. Initiation of CFTR modulator within previous 8 weeks OR unstable changes in weight and lung function due to CFTR modulator use
13. Actively trying to gain or lose weight
14. Any food allergies or intolerances that cannot be accommodated
15. Any medical condition deemed by the a study physician or PI that may preclude completion of the study or interfere with primary end points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in acute insulin response to arginine (AIRarg) from baseline | Baseline and 8 weeks post intervention
  Participants will undergo a Glucose-Potentiated Arginine Stimulation (GPA) Test after a 10-12 hour overnight fast to measure acute insulin (AIRarg) responses during a 230 and 340 mg/dl glucose clamp. This test will measure changes in beta cell secretory capacity.
Change in acute C-peptide (ACRarg) from baseline | Baseline and 8 weeks post intervention
  Participants will undergo a Glucose-Potentiated Arginine Stimulation (GPA) Test after a 10-12 hour overnight fast to measure acute C-peptide (ACRarg) responses during a 230 and 340 mg/dl glucose clamp. This test will measure changes in beta cell secretory capacity.
Change in visceral adipose tissue from baseline | Baseline and 8 weeks post intervention
  Dual energy X-ray absorptiometry (DEXA)-derived measurement of visceral adipose tissue (VAT) will be assessed with a GE Lunar iDXA machine. This will enable assessment of changes in body composition over the study.
Change in fasted plasma Eh[CySS] from baseline | Baseline and 8 weeks post intervention
  Change in plasma Cysteine/Cystine Redox Potential (Eh[CySS]) will be measured.

SECONDARY OUTCOMES:
Change in Gastrointestinal Symptom Rating Scale (GSRS) scale | Baseline and 8 weeks post intervention
  The GSRS is a 15 items combine into five symptom clusters: Reflux, Abdominal pain, Indigestion, Diarrhea and Constipation.
  Possible score range is 0-7, with 7 being the worst and 0 being the best (no symptoms).
Change in hepatic and pancreatic fat volume | Baseline and 8 weeks post intervention
  Dual energy X-ray absorptiometry (DEXA)-derived measurement of visceral adipose tissue (VAT) for hepatic and pancreatic fat volume. Will be assessed with a GE Lunar iDXA machine.
Change in fasted plasma Eh[GSSG] | Baseline and 8 weeks post intervention
  Change in plasma glutathione disulfide (GSSG) (Eh[CySS]) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Alvarez, PhD, RD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Actual clinical study data in raw and summary form, with protected health information removed, as well as access to the study database, will be available for reference of qualified professional colleagues and auditors up to 10 years after study publication. With appropriate subject informed consent, clinical and research data obtained from this study will be deposited into the Georgia CF Data Warehouse of the NDDK P30-supported Georgia Cystic Fibrosis Clinical and Translational Core Center.
Supporting Information: Study Protocol
Time Frame: After final publication date
Access Criteria: Qualified researchers for analyses of original study endpoints not pre-specified as primary, secondary, or exploratory that contact the investigators.

REFERENCES:
- [Derived] Zaveri S, Stecenko A, Hunt WR, Goss A, Sharma P, Hartman TJ, Easley K, Chandler JD, Burley TM, Driggers C, Ciccarella A, Zhou H, Narlow K, Ziegler TR, Daley T, Vellanki P, Alvarez J. Low-added sugar dietary intervention study to mitigate glucose intolerance and improve body composition in adults with cystic fibrosis: a protocol of a double-blind, randomised study. BMJ Open. 2024 Dec 26;14(12):e092503. doi: 10.1136/bmjopen-2024-092503. PMID 39725418